CLINICAL TRIAL: NCT00842036
Title: CRAFT Behavior Therapy Phase 2 Study: Treatment Entry Component
Brief Title: CRAFT Behavior Therapy: Treatment Entry Component
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Responsible Party: Kimberly C. Kirby, Ph.D., Principal Investigator, Treatment Research Institute
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0406; 5R01DA018696 (NIH)
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Drug Addiction; Stimulant Dependence; Opiate Dependence; Alcohol Dependence; Substance Abuse
Keywords: Family Therapy; Relationship Dysfunction; Family Dysfunction; Family Relations; Stimulant Dependence; Opiate Dependence; Alcohol Dependence; Behavior Therapy; Drug Treatment; Substance Abuse; Drug Addiction
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ANft (Active Comparator): 12- step Al/Nar-Anon Facilitation
  Interventions: Behavioral: 12- step Al/Nar- Anon Facilitation
- TEnT (Experimental): Treatment Entry Training
  Interventions: Behavioral: Treatment Entry Training
- CRAFT (Experimental): Community Reinforcement and Family Training
  Interventions: Behavioral: Community Reinforcement and Family Training

INTERVENTIONS:
Behavioral: Community Reinforcement and Family Training — Community Reinforcement and Family Training (CRAFT) is an intervention designed for the concerned significant other (CSO) of a drug or alcohol using loved one. The CRAFT intervention consists of approximately 12 sessions lasting 45-60 minutes. The goal of the CRAFT intervention is to train the CSO in new ways to interact with the person of concern (PC). There are four components that the CSO is trained on which include awareness training, community reinforcement training, treatment entry training, and CSO mood enhancement.
  Arms: CRAFT
Behavioral: Treatment Entry Training — Treatment Entry Training (TEnT) is a component of the Community Reinforcement and Family Training intervention and it is currently under investigation to determine if it is sufficient to produce the primary and most consistent outcome of CRAFT- treatment entry of the drug user. The intervention will consist of a minimum of 4 sessions and a maximum of 6 sessions that are each 45-60 minutes long. TEnT will include awareness training, safety training, and the Treatment Entry Training component of CRAFT.
  Arms: TEnT
Behavioral: 12- step Al/Nar- Anon Facilitation — The underlying philosophy of the 12- step approach for concerned significant others (CSO) is that the CSO is powerless to control the drinker/drug user and must detach, focusing instead on accepting the situation and on strengthening his or her mental health. Eight content areas are discussed with the CSO over the course of the intervention. There will be a minimum of 8 sessions and a maximum of 12 sessions that are each 45-60 minutes long.
  Arms: ANft

SUMMARY:
This research compares the benefits of the original treatment, Community Reinforcement and Family Training (CRAFT), with the Treatment Entry Training (TEnT) component of CRAFT to determine if TEnt alone can produce the primary outcome of CRAFT -- treatment entry of the drug user. We also look at the impact on the well-being of the concerned significant other and the drug use of their loved one.

DETAILED DESCRIPTION:
The consequences of drug abuse are not limited to drug users; they also extend to their families and concerned significant others (CSOs). Research shows that CSOs of drug users have increased prevalence of illness, domestic violence, and problems in mood and functioning. Because CSOs are troubled by the negative effects of drug use on the drug user and themselves, they may be a social community that is particularly invested in learning ways to positively influence the drug user.

We compare the benefits of the original treatment, Community Reinforcement and Family Training (CRAFT), with the Treatment Entry Training (TEnT) component of CRAFT to see if the TEnt is sufficient to produce the primary and most consistent outcome of CRAFT -- treatment entry of the drug user.

ELIGIBILITY:
Inclusion Criteria:

* Concerned Significant Other (CSO) and Person of Concern (PC) over 18 years of age
* is a family member (such as a close relative, spouse, intimate partner), roommate or significant other who is concerned about a PC
* reports that the PC has a pattern of drug or alcohol use that meets the criterion for abuse or dependence on stimulants, opiates, or alcohol according to DSM-IV-TR
* reports that the PC is not currently in treatment and has not received treatment during the past 6 weeks (other than detoxification)
* reports having been in the relationship with the identified PC for at least 3 months
* reports contact with the identified PC on at least 12 of the past 30 days with no planned change in the amount of contact in the next 10 months
* provides evidence that the PC has refused to seek treatment when CSO asked

Exclusion Criteria:

* does not demonstrate complete understanding of their participation by reading the consent form and passing a consent quiz that tests comprehension of the basic elements of informed consent and requirements of the protocol, or does not agree to participate by signing an informed consent
* declines to: provide valid locator information, allow videotaped sessions, and/or participate in follow-ups
* CSO has a drug abuse problem themselves as determined through clinical assessment and DSM-IV-TR criteria
* is not able to comprehend the content in the self-report materials (written at about 6th grade reading level)
* reports that the PC behaves in a manner consistent with an unremitting psychosis or another psychiatric disorder (e.g., significant developmental delay) that would contraindicate the planned CRAFT intervention
* intends to receive more than 6 hours of individual counseling focusing on the PC's addiction for the 6 months after they are enrolled in the study
* PC has a recent history of severe domestic violence (e.g., the PC has committed criminal assault during the past 2 years, or has a history of severe violence involving a weapon or resulting in hospitalization
* has an immediate family member, friend, roommate, co-worker, or other person who has already enrolled in the study and his/her participation is not likely to be independent of the initially enrolled CSO's participation
* fails to complete 2 sessions with a family trainer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Treatment entry of the drug user | This may occur at any point throughout the participants' involvement in the study

SECONDARY OUTCOMES:
Reduction in drug use | 2 month, 4 month, 6 month, and 9 month assessments
Improvements in mood and functioning | 2 month, 4 month, 6 month, and 9 month assessments

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly C Kirby, Ph.D., Principal Investigator — Treatment Research Institute
Locations (1):
- TRI South Street, Philadelphia, Pennsylvania, United States